CLINICAL TRIAL: NCT06827691
Title: Heat Therapy for People with Peripheral Artery Disease: a Randomised Wait-List Controlled Feasibility Trial.
Brief Title: Heat Therapy and Peripheral Artery Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EthOS: 71125
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Health; Vascular Function; Intermittent Claudication; Peripheral Vascular Diseases
Keywords: heat therapy; cardiovascular health; endothelial function; heat intervention
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Randomised wait-list controlled feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait-list control (No Intervention): Usual care 8 weeks
- Heat Therapy Intervention (Active Comparator): Heat therapy intervention through water submersion in a hot tub at ~40°C.
  Interventions: Other: Heat Therapy Intervention

INTERVENTIONS:
Other: Heat Therapy Intervention — Heat Therapy Intervention of shoulder depth submersion in a 40°C hot tub.
  Arms: Heat Therapy Intervention

SUMMARY:
The purpose of the study is to assess the efficacy of a novel 8 week heat therapy intervention in intermittent claudication compared to usual care controls. Participants will be enrolled on a wait-list control randomised trial testing physiological, mechanistic, and health related outcome measures.

DETAILED DESCRIPTION:
70 participants with PAD will be randomised into one of two groups: either wait-list controls (usual care) or heat therapy intervention. The 8 week heat therapy intervention will consist of shoulder depth submersion in a hot tub at ~40°C for three times a week. Time for heating will be graded with aim of ~60 minutes submersion time by the end of the intervention. After 8 weeks the wait-list control group will then enrol onto the heat intervention and heat therapy participants will go back to usual care. The primary outcome measure for the study is improvement in maximum walking distance, pain free walking, and time to onset claudication. This will be measured via a graded exercise test. Secondary outcomes include Quality of life as measured by generic and vascular specific questionnaires (SF-36,VascuQoL and EQ-5D-5L), vascular health measured using ABPI, blood pressure, FMD, PWV, and markers of inflammation, oxidative stress, angiogenesis and vascular remodelling will be assessed from blood samples. All aforementioned outcome measures will be taken at baseline, 8 weeks, and 16 weeks. Physical activity behaviour (measured with an accelerometer) will be monitored 7 days prior to the beginning of the study, 7 days prior heat intervention, and 7 days after heat intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Aged > 18 years

  * ABPI < 0.9 at rest or a drop of 20mmHG after exercise testing
  * Diagnosed with IC
  * Able to walk unaided
  * English-speaking and able to follow instructions
  * No previous history of heat syncope
  * Post-Menopausal or not on hormone therapy
  * Able to provide informed consent

Exclusion Criteria:

* • Walking impairment for a reason other than PAD

  * Critical limb ischaemia/rest pain
  * Asymptomatic PAD
  * Active cancer treatment
  * Clinically diagnosed diabetes or those with peripheral neuropathy
  * Recent / frequent heat exposure (e.g., sauna or hot tubs).
  * severe aortic stenosis, unstable angina, recent MI, stroke or TIA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Walking Distance | Baseline to 8 weeks to 16 weeks
  Maximal walking distance a participant can walk, through a graded treadmill test.
Pain Free Walking Distance | Baseline to 8 weeks to 16 weeks
  Maximum distance participant can walk without pain (IC)
Time for Onset of Claudication | Baseline to 8 weeks to 16 weeks
  Amount of time able to walk pain free before reaching claudication

SECONDARY OUTCOMES:
VascuQoL-6 | Baseline to 8 weeks to 16 weeks
  Quality of life was assessed using the Vascular Quality of Life Questionnaire (VacQoL), a disease-specific instrument comprised of 25 items rated on a 7-point Likert scale. When scored as a mean across items, the VacQoL has a range from 1 to 7, where 1 indicates the poorest quality of life and 7 the best. Alternatively, when summed, the total score ranges from 25 (worst) to 175 (best).
SF-36 | Baseline to 8 weeks to 16 weeks
  The Short Form 36 Health Survey Questionnaire (SF-36) is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions.
EQ-5D-5L | Baseline to 8 weeks to 16 weeks
  The EQ-5D-5L is a brief, multi-attribute, generic, health status measure composed of 5 questions with Likert response options (descriptive system) and a visual analogue scale. The latter asks patients to rate their own health from 0 to 100 (the worst and best imaginable health, respectively).
Markers of Inflammation | Baseline to 8 weeks to 16 weeks
  Investigators will compare blood sample measures of TNF-α, CRP, MCP-1, IL-1Ra, IL-4, IL-6, IL-8, IL-10, and eHSP70.
Markers of Vascular Remodelling | Baseline to 8 weeks to 16 weeks
  Investigators will compare blood sample measures of HIF-1α, VEGF, endothelin-1, MMP-9, MMP-10 and nitrite.
Tissue Oxygenation | Baseline to 8 weeks to 16 weeks
  Superficial tissue oxygen saturation and muscle oxygen consumption will be measured throughout the protocol by a NIRS probe placed on the skin surface of the medial gastrocnemius on the most affected leg. Measurements will be recorded during the graded treadmill test.
Vascular Ultrasound Imaging | Baseline to 8 weeks to 16 weeks
  Vascular ultrasound images of the carotid, brachial and superficial femoral artery will be obtained using a high-resolution duplex machine (Terason, Burlington, MA) and subsequently used to calculate wall thickness, changes in arterial blood flow and shear stress.
Flow-Mediated Dilation | Baseline to 8 weeks to 16 weeks
  Flow-mediated dilation (FMD) of the brachial artery will be measured after 10 min of supine rest via reactive hyperemia in response to transient ischemia of the lower arm according to international guidelines.
Ankle-Brachial Pressure Index | Baseline to 8 weeks to 16 weeks
  Ankle brachial pressure index (ABPI): ABPI will be determined at rest and following a treadmill test by using standardised methodologies
Blood Pressure | Baseline to 8 weeks to 16 weeks
  Following a 10-minute period of supine rest in a quiet room, blood pressure will be measured (in duplicate) using an automated sphygmomanometer.
Pulse Wave Velocity and Pulse Wave Analysis | Baseline to 8 weeks to 16 weeks
  Pulse wave velocity will be measured using central (carotid-femoral) and peripheral (carotid-radial) via a handheld tonometer following standard guidelines. This will be used with a SphygmoCor XCEL.
Physical Activity Levels | 7 days prior trial, 7 days prior heat intervention, 7 days after heat intervention, 7 days post trial.
  Physical activity will be measured using a wrist-worn accelerometer. Physical activity will be monitored for 7 days at a time. This including 7 days pre-trial, 7 days pre heat intervention, 7 days post heat intervention, and 7 days post trial (Dependent on what group randomisation was first).

OTHER OUTCOMES:
Intervention feasibility assessed via recruitment rate | through study completion, an average of 1 year
  The investigators will record the number of eligible participants, as well as the number who enrol onto the study.
Intervention feasibility assessed via protocol adherence | through study completion, an average of 1 year
  The investigators will examine adherence on visits to the lab for the heat therapy intervention. I.e. How many sessions were completed throughout the 8 weeks.
Intervention acceptability via workshop interviews | through study completion, an average of 1 year
  Workshop interviews will be held between an investigator and participants who has either completed the intervention, withdrawn or declined participation, to ask questions regarding the intervention protocol.
Intervention feasibility via participant comfort | through study completion, an average of 1 year
  The investigators will examine participant thermal comfort/discomfort throughout each intervention day. This will be done through recording of time spent in tub and thermal comfort scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Metropolitan University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No